CLINICAL TRIAL: NCT01670071
Title: A Randomized, Open-Label, Study To Evaluate The Effect of Oral Paliperidone Extended-Release and Oral Risperidone Immediate-Release on Selected Cognitive Domains in Clinically Stable Subjects With Schizophrenia
Brief Title: A Study to Evaluate the Effect of Oral Paliperidone Extended-Release and Oral Risperidone Immediate-Release on Cognitive Function in Clinically Stable Patients With Schizophrenia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated due to insufficient sample size and protocol compliance issue.
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100817; R076477SCH4066 (Other: Johnson & Johnson Taiwan Ltd)
Record Dates: First submitted 2012-08-17; First posted 2012-08-21 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone; Risperidone; Paliperidone extended-release (ER); Risperidone immediate-release (IR)
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paliperidone extended-release (Experimental)
  Interventions: Drug: Paliperidone extended-release
- Risperidone immediate-release (Active Comparator)
  Interventions: Drug: Risperidone immediate-release

INTERVENTIONS:
Drug: Paliperidone extended-release — Patients will receive 6 mg to 12 mg of paliperidone extended-release tablet once daily orally.
  Other Names: Paliperidone
  Arms: Paliperidone extended-release
Drug: Risperidone immediate-release — Patients will receive 3 mg to 7 mg of risperidone immediate-release tablet orally.
  Other Names: Risperidone IR
  Arms: Risperidone immediate-release

SUMMARY:
The purpose of this study is to compare the effect of oral paliperidone extended-release and oral risperidone immediate-release on cognitive function, especially the category fluency of Cognitive Abilities Screening Instrument, Chinese version (CASI C-2.0), in patients with an established diagnosis of schizophrenia.

DETAILED DESCRIPTION:
This is a 28-week, randomized (the study medication is assigned by chance), open-label (all people know the identity of the intervention), active-controlled (patients are assigned to either a recognized effective treatment or the study medication) comparative study. All patients will enter a run-in period to receive a stable therapeutic dose of oral risperidone immediate-release for at least 4 weeks. After the 4-week run-in period, patients will be randomly assigned to either remain on oral risperidone immediate-release (IR) or to receive a therapeutic dose of oral paliperidone extended-release (ER) and patients will be prospectively followed for a 24-week treatment phase. The treatment phase is composed of a 4-week flexible dose period followed by a 20-week stable dose period. During the 4-week flexible dose period, the dose of paliperidone ER or risperidone IR may be increased or decreased for each patient if clinically indicated (eg, significant side effects emerge or there is evidence of a lack of efficacy). At the end of 4-week flexible dose period, the final dose should be maintained for the 20-week fixed-dose period. Efficacy and safety will be assessed at baseline (Week 0) and Weeks 4, 12, and 24.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with schizophrenia
* Cognitive abilities screening instrument C-2.0 total score between 50 and 85 (inclusive) at baseline
* Baseline positive and negative syndrome scale score between 60 and 85 (inclusive)
* Clinical global impression-severity change less than or equal to 1 in the month prior to randomization
* Patients on a stable therapeutic dose of oral risperidone IR (between 3-6 mg/day) for at least 4 weeks prior to randomization

Exclusion Criteria:

* Treatment refractory patients, defined as failure of more than or equal to 2 adequate trials of second generation antipsychotic treatment for schizophrenia
* History of neuroleptic malignant syndrome
* Allergy or hypersensitivity to risperidone or paliperidone, or to any of the excipients of oral risperidone IR or paliperidone ER tablets
* Participants who have taken paliperidone ER in the past
* Participants who have been treated with clozapine or any long-acting injectable (depot) antipsychotic within 3 months before randomization

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in category fluency score of cognitive function scale (Cognitive Abilities Screening Instrument, Chinese version [CASI C-2.0]) from baseline to Week 24 | Baseline (Week 0), Week 4, Week 12 and Week 24
  CASI C-2.0 will be used to measure patient's cognitive ability. The range of CASI score is 0 to 100 (a higher score indicating better performance and is influenced by patient's educational level). The CASI C-2.0 provides quantitative assessment on 9 cognitive domains and 20 questions, including attention, concentration, orientation, short-term memory, long-term memory, language abilities, visual construction, category fluency, abstraction, and judgment.

SECONDARY OUTCOMES:
Change from baseline to Week 24 in score of Modified Wisconsin Card Sorting Test (MWCST) short version | Baseline, Week 4, Week 12 and Week 24
  The WCST was developed to assess abstract reasoning and ability to shift cognitive strategies in response to environmental changes. The materials consist of a pack of 4 stimulus cards and 48 response cards which are devised so that each card contains from 1 to 4 identical figures of a single color. Individually administered, it requires the patient to sort the cards according to different principles (ie, by color, form, or number). As the test progresses, there are unannounced shifts in the sorting principle which require the patient to alter his or her approach.
Change from baseline in score of Continuous Performance Test (CPT) | Baseline, Week 4, Week 12 and Week 24
  CPT is an attention test. Response patterns on the CPT II is used as an aid in monitoring treatment effectiveness. For example, some response patterns suggest inattentiveness or impulsivity, while other response patterns may indicate activation/arousal problems or difficulties maintaining vigilance.
Change from baseline in score of Personal and Social Performance (PSP) scale | Baseline, Week 4, Week 12 and Week 24
  The PSP is a clinician-rated instrument providing an overall rating of personal and social functioning in subjects with schizophrenia on a scale of 1-100. Four domains of functioning are considered in the rating: 1) socially useful activities, including work and study, 2) personal and social relationships, 3) self-care, and 4) disturbing and aggressive behavior.
Change from baseline in score of Positive and Negative Syndrome Scale (PANSS) | Baseline, Week 4, Week 12 and Week 24
  The PANSS is a medical scale used for measuring symptom severity of patients with schizophrenia. The neuropsychiatric symptoms of schizophrenia will be assessed using the 30-item PANSS scale, which provides a total score (sum of the scores of all 30 items). Each scale is rated 1 (absent) to 7 (extreme).
Change from baseline in score of Clinical Global Impression-severity (CGI-S) scale | Baseline, Week 4, Week 12 and Week 24
  The CGI-S rating scale is used to rate the severity of a patient's psychotic condition on a 7-point scale ranging from 1 (not ill) to 7 (extremely severe). This scale permits a global evaluation of the patient's condition at a given time.
Change from baseline in score of Medication Satisfaction Questionnaire (MSQ) | Baseline, Week 4, Week 12 and Week 24
  MSQ is designed to assess treatment satisfaction among patients with schizophrenia. It consists of 1 question: "Overall, how satisfied are you with your current antipsychotic medication(s)?" with responses assessed on a 7-point scale rated as follows: 1=extremely dissatisfied, 2=very dissatisfied, 3=somewhat dissatisfied, 4=neither satisfied nor dissatisfied, 5=somewhat satisfied, 6=very satisfied, and 7=extremely satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan Ltd Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd
Locations (3):
- Taiwan (3):
  - Bali Township, Taipei County
  - Hualien City
  - Kaohsiung City

REFERENCES:
- See also: Paliperidone ER and oral risperidone - A 6-month prospective pilot RCT, exploring differential effects on cognitive domains in patients with schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=3485&filename=CR100817_CSR.pdf